CLINICAL TRIAL: NCT07336810
Title: Effect of Whole-Body Vibration Versus Neuro Muscular Electrical Stimulation on Patients With Intensive Care Acquired Weakness
Brief Title: Whole-Body Vibration Versus Neuro Muscular Electrical Stimulation on Patients With ICU Acquired Weakness
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, AHMED REFAAT ABD EL AZIZ TAHA MALIK, Principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/005115; P.T.REC/012/005115 (Other: Cairo University)
Record Dates: First submitted 2025-11-24; First posted 2026-01-13 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Muscle Weakness | Patient; Intensive Care (ICU) Myopathy; Intensive Care (ICU)
Keywords: Intensive Care Unit Acquired Weakness; NEURO MUSCULAR ELECTRICAL STIMULATION
MeSH Terms: conditions — Muscular Diseases

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A ( Whole body vibration) (Active Comparator): each patient who will practice Whole body vibration for two weeks twice daily in addition to their plan of treatment.
  Interventions: Device: whole body VIBRATION Viberation
- Group B (NEURO MUSCULAR ELECTRICAL STIMULATION B ) (Active Comparator): Each patient will receive neuromuscular electrical stimulation for two weeks, twice daily, in addition to their plan of treatment
  Interventions: Device: Neuro muscular electrical stimulation

INTERVENTIONS:
Device: whole body VIBRATION Viberation — Whole body vibration will be applied twice daily for two weeks. The patients will be in the supine position during the entire intervention, and no changes in body position will take place to avoid any influence on hemodynamic parameters and vital signs. Following baseline measurements, patients will be mobilized passively for 6 minutes as a warm-up. whole body vibration treatment will be initiated, consisting of a vibration plate device will placed under the patient's feet, with resistance to the end of the bed. The patient's hips and knees will be flexed at about 20°. An elastic strip will provide pressure on the knees, pushing the patient's feet against the vibration device. Whole body vibration sessions took 15 minutes, with 9 minutes of clear vibration time. The vibration frequency will be 25 HZ and the amplitude of 2 mm
  Arms: Group A ( Whole body vibration)
Device: Neuro muscular electrical stimulation — Neuromuscular electrical stimulation will be applied twice daily for two weeks. 20 min per muscle group bilaterally on eight different muscle groups (triceps surau (calf muscle), Quadriceps, Hamstring, biceps brachii, triceps brachii, wrist extensors and shoulder abductors). We will never stimulate counteracting muscle groups at the same time. Electrical impulses of 350 μs duration will be applied at a frequency of 50 Hz. Electrical current will be increased until muscle contraction can be visible or palpable, which can be tolerable and does not cause pain or discomfort, and then it will be maintained at this level for the remainder of the session.
  Arms: Group B (NEURO MUSCULAR ELECTRICAL STIMULATION B )

SUMMARY:
Purpose: to investigate the effect of Whole-body vibration versus neuro-muscular electrical stimulation on patients with intensive care-acquired weakness. Methods: Sixty patients with Intensive Care Unit-acquired weakness (ICU AW) from both genders will be recruited and randomly assigned into two groups, Group A and Group B. Group A will include 30 patients who will practice Whole body vibration for two weeks twice daily in addition to their plan of treatment. Group B will include 30 patients who will receive neuromuscular electrical stimulation for two weeks, twice daily, in addition to their plan of treatment. All patients will be evaluated pre- and post-treatment for the MRC score, creatine phosphokinase, and total muscle strength and skeletal muscle thickness

DETAILED DESCRIPTION:
A) Procedure for evaluation:

The practical section of the study will be undertaken in 2 weeks (two sessions per day). Measurements will be taken before the start of the training program then after the end of the 2-week training program in the following manner:

1. Manual muscle test (MMT) and medical research council score (MRC): will be used to assess muscle strength.
2. Laboratory investigations for CPK: Blood serum samples will be collected. For each sample, 5 mL of blood will be drawn for laboratory analyses to detect damage in skeletal muscle.
3. Strength Testing with Dynamometry: A Handheld Dynamometer will be used to assess the skeletal muscle strength objectively.
4. Skeletal muscle ultrasonography: will be used to assess the size and thickness of muscles.

B) Training procedures:

All patients in both groups will receive their plan of treatment in addition to the training program for each group as follows:

Group (A) patients in this group will participate in Whole Body Vibration (WBV) training for 2 weeks, two sessions per day (total 14 sessions) in addition to their plan of treatment.

Group (B) patients in this group will participate in neuromuscular electrical stimulation (NMES) training for 2 weeks, two sessions per day ( total 14 sessions), in addition to their plan of treatment.

C) The statistical analysis will be conducted by using the SPSS statistical package program version 25 for Windows (SPSS, Inc., Chicago, IL). Quantitative descriptive statistics data, including the mean and standard deviation, will be used to describe the data. Multivariate analysis of variance (MANOVA) will be used to compare the tested major dependent variables of interest. A mixed-design 2 x 2 MANOVA test will be used to detect within-group changes and between-group differences. The Bonferroni correction test will be used for pairwise comparison within and between groups of the tested dependent variables, whose P-value will be significant from the MANOVA test. The significance level for all statistical analyses will be set at p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* ICU patients who were aged ≥ 18 and <65.
* Sepsis-related Organ Failure assessments (SOFA) score ≥ 9 within the first 72 h after ICU admission.
* Patients with no central and peripheral nervous system injury.
* Expected to be treated in the ICU for more than 1 week.
* Medical Research Council (MRC) sum score of less than 36/60.
* Dominant-hand handgrip dynamometry scores of less than 11 kg (interquartile range (IQR) 10-40) in males and less than 7 kg (IQR 0-7.3) in females

Exclusion Criteria:

* Patients with comorbidities interfering with or compromising the training, like cardiac arrhythmia, pericardial effusion, congestive heart failure, or unstable acute coronary syndrome.
* Patients are hemodynamically unstable.
* Patients who had a major neurological deficit (upper motor neuron lesion).
* Age < 18 years and more than 65.
* Implanted pacemaker or defibrillator.
* Pregnancy.
* Unhealed fractures or recently attached implants in the body region to be stimulated.
* Acute venous thrombosis.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2026-01-10 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Manual muscle test (MMT) | At baseline and post two weeks
  manual muscle testing will be assessed bilaterally, including tibialis anterior, triceps surau, Quadriceps, hamstrings, biceps brachii, triceps brachii, and wrist extensors. these muscles will be assessed in 5 grades of muscle testing, where grade zero means no contraction and grade five means active movement through the full range of motion against full applied resistance against gravity
Medical Research Council (MRC) | At baseline and post two weeks
  The MRC scale will be used for early detection of muscle strength, as it has a score ranging from 0 to 60, where < 48 means significant weakness
change of Creatine phosphokinase (CPK-MM) | change from baseline CPK-MM level at 2 weeks
  The Beckman Unicel DxC800 method will be used for measuring serum CPK-MM
muscle strength | At baseline and post two weeks
  Handheld dynamometry (HHD) will be used to measure the muscle strength of the selected muscles by quantifying the force generated when a person pushes or pulls against a stationary device.
Muscle thickness | at baseline and post 2 weeks
  Skeletal muscle ultrasonography will be used to assess muscle thickness

CONTACTS AND LOCATIONS:
Overall Officials: Heba A. Abd El Ghafar,, A. Professor, Study Director — Cairo University
Locations (1):
- critical care department (DR. Sherief Mokhtar unit) in kasr Al-Ainy medical school, Cairo, Egypt., Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No